CLINICAL TRIAL: NCT01525329
Title: Combination Therapy With 5-Fluorouracil and Photodynamic Therapy for the Treatment of Post-transplant Premalignant Skin Disease
Brief Title: Combination Therapy With 5-Fluorouracil and Photodynamic Therapy in Post-transplant Premalignant Skin Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: study drug no longer available in the United States
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Maytin, MD, PhD, Section Head, Molecular Dermatology; Chairman, Dermatology Research Committee, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-1050; 1R21CA156227-01A1 (NIH)
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Actinic Keratosis; Organ or Tissue Transplant; Complications
Keywords: Actinic Keratosis; Photodynamic Therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solid Organ Transplant with AKs (Experimental): Patients who have undergone kidney or liver transplant within 2 years and have at least 4 premalignant skin lesions on the face, ears, scalp, forearms and/or dorsal hands. Patients will serve as their own control, and one side of the body will be randomized to either 5-FU plus PDT, and the other will receive PDT alone.
  Interventions: Drug: 5-Fluorouracil
- Actinic Keratoses (Active Comparator): Patients with at least 4 actinic keratoses on the face, ears, scalp, forearms and/or dorsal hands. Patients will serve as their own control, and one side of the body will be randomized to either 5-FU plus PDT, and the other will receive PDT alone.
  Interventions: Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: 5-Fluorouracil — All patients will receive one cream, 5-Fluorouracil, and will be instructed to apply the cream according to the randomization schema to AKs on either the right or left side of the face/scalp once a day for 6 days prior to PDT. A baseline measurement of the tumor's ability to produce PpIX will be done by applying methyl-aminolevulinic acid (Metvixia® topical cream) to the selected AKs and using the Aurora© dosimeter. Prior to Metvixia, and again 3 hours after application, surface measurements of the PpIX fluorescence will be taken. Then, the two largest precancer lesions (one on the left side, one on the right side) will be biopsied under local anesthesia, followed by red light PDT (lasting ~8 minutes). The biopsy sites will be shielded from the light with a circular spot bandage.
  Other Names: Fluorouracil Cream, USP 5%; 5-FU

SUMMARY:
This randomized, intra-patient comparative study is designed to investigate the combination regimen of 5-fluorouracil cream (5FU) and Photodynamic Therapy (PDT), versus PDT alone, for its ability to generate significantly elevated levels of the target photosensitizer, protoporphyrin IX (PpIX), in lesions of actinic keratoses (AKs) and to more effectively treat and prevent recurrence of AKs. The target population comprises patients with solid organ transplants (renal, hepatic), as well as normal (immunocompetent) subjects to control for possible influences of immunosuppression.

DETAILED DESCRIPTION:
This clinical trial will test a new combination of 5-fluorouracil cream (5FU) and methylaminolevulinate photodynamic therapy (MAL-PDT), versus MAL-PDT alone, as treatment for actinic keratoses (AKs) in immunosuppressed organ transplant recipients (OTRs) and an immunocompetent control group. Objectives: 1) Determine whether topical pretreatment with 5-FU selectively increases the amount of photosensitizer (PpIX) produced within AK lesions, relative to non-pretreated lesions. 2) Determine whether the combination treatment improves lesion resolution and reduces the incidence of new AKs. 3) Determine whether biomarkers in tissue and blood are predictive of patient responsiveness to 5FU (PpIX induction, new lesion incidence, and clinical toxicity).

We plan to enroll 20 organ transplant recipients and 20 normal patients, with AKs on face, scalp, ears, forearms or back of the hand through Dermatology and Transplant Clinic at Cleveland Clinic. Women of childbearing age must use contraception and have a negative pregnancy test.

Study participants will apply 5FU daily for 6 days; MAL/PDT is administered on 7th day. PpIX will be measured in lesions using a noninvasive dosimeter. Biopsies will be taken from selected lesions, and AKs will be photographed. Participants will be asked to complete a questionnaire to document adverse events. Patients are evaluated at day 14, and months 3, 6, 9, 12, to document AK clearance and new lesion appearance.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* At least four (4) actinic keratoses, located on face, ears, scalp, forearms and/or dorsal hands. - Patients in the solid organ transplant arm of the study must have had either a kidney or liver transplant, and the transplantation surgery must have occurred at least 2 years prior to enrollment.

Exclusion Criteria:

* Pregnant or nursing
* Currently participating in another clinical trial
* Using any topical treatment for their actinic keratoses
* Currently being treated for other cancers with medical or radiation therapy
* Patients with a known hypersensitivity to 5-aminolevulinic acid, 5-fluorouracil or any component of the study material
* Patients with a history of a photosensitivity disease, including porphyria cutanea tarda

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Maytin, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual participant data with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Solid Organ Transplant With AKs: Patients who underwent kidney or liver transplant within 2 years, and with at least 4 premalignant skin lesions on face, ears, scalp, forearms or dorsal hands. Patients will serve as their own control; one side of the body will be randomized to 5-FU plus PDT, and the other to PDT alone.
  All patients will receive one cream, 5-Fluorouracil (5FU), and will apply it to the AKs on either the right or left side of the face/scalp (per randomization scheme), once daily for 6 d prior to PDT. The ability of AKs to produce PpIX will be measured at baseline by applying methyl-aminolevulinate (Metvixia® topical cream) to the selected AKs using a fluorescence dosimeter. Prior to Metvixia, and again 3 hours after application, surface measurements of PpIX fluorescence will be taken. Then the two largest lesions (one on the left, one on the right) will be biopsied under local anesthesia, followed by red light PDT (lasting ~8 minutes). Biopsy sites will be shielded from light with a spot bandage.
- Actinic Keratoses: Patients with at least 4 actinic keratoses on the face, ears, scalp, forearms and/or dorsal hands. Patients will serve as their own control, and one side of the body will be randomized to either 5-FU plus PDT, and the other will receive PDT alone.
  All patients will receive one cream, 5-Fluorouracil (5FU), and will apply it to the AKs on either the right or left side of the face/scalp (per randomization scheme), once daily for 6 d prior to PDT. The ability of AKs to produce PpIX will be measured at baseline by applying methyl-aminolevulinate (Metvixia® topical cream) to the selected AKs using a fluorescence dosimeter. Prior to Metvixia, and again 3 hours after application, surface measurements of PpIX fluorescence will be taken. Then the two largest lesions (one on the left, one on the right) will be biopsied under local anesthesia, followed by red light PDT (lasting ~8 minutes). Biopsy sites will be shielded from light with a spot bandage.
Period: Overall Study
Arm/Group | Solid Organ Transplant With AKs | Actinic Keratoses
Started | 4 | 14
Completed | 4 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Solid Organ Transplant With AKs: Patients who underwent kidney or liver transplant within 2 years, and with at least 4 premalignant skin lesions on face, ears, scalp, forearms or dorsal hands. Patients will serve as their own control; one side of the body will be randomized to 5-FU plus PDT, and the other to PDT alone.
- Total: Total of all reporting groups
Arm/Group | Solid Organ Transplant With AKs | Actinic Keratoses | Total
Number analyzed (Participants) | 4 | 14 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 10 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 11 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 14 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Accumulation of Porphyrin (PpIX)
Description: The primary endpoint of this study will be the accumulation of PpIX at 3 h after MAL application (measured noninvasively, in each treated region).
  (Region refers to the half-face or half-scalp area treated with PDT monotherapy, or the contralateral area treated with the 5-FU/PDT combination regimen).
Time Frame: Day 7 of the study
Measure: Mean (95% Confidence Interval); unit: Change in PpIX signal (arbitrary units)
Groups:
- Transplant With AKs; 5FU + PDT: Patient with solid organ transplant: half of body receiving combination therapy
- Transplant With AKs; PDT Only: Patient with solid organ transplant: half of body receiving PDT alone
- Normals With AKs; 5FU + PDT: Patient without any organ transplant: half of body receiving combination therapy
- Normals With AKs; PDT Only: Patient without any organ transplant: half of body receiving PDT alone
Arm/Group | Transplant With AKs; 5FU + PDT | Transplant With AKs; PDT Only | Normals With AKs; 5FU + PDT | Normals With AKs; PDT Only
Number analyzed (Participants) | 4 | 4 | 14 | 14
Change in PpIX signal (arbitrary units) | 101.8 [45.1 to 158.4] | 48.0 [-2.0 to 98.0] | 84.3 [60.6 to 108.0] | 38.4 [15.1 to 61.6]
Statistical Analysis 1: Comparison: Transplant With AKs; 5FU + PDT vs Transplant With AKs; PDT Only; Test type: Superiority or Other; p < 0.007, t-test, 2 sided
Statistical Analysis 2: Comparison: Normals With AKs; 5FU + PDT vs Normals With AKs; PDT Only; Test type: Superiority or Other; p = 0.080, t-test, 2 sided

2. Secondary Outcome: Actinic Keratosis (AK) Clearance
Description: Rate of AK clearance (Analyzed by linear mixed-effect model)
Time Frame: AK counts, over a 12-month period
Measure: Mean (95% Confidence Interval); unit: CR (% reduction)
Arm/Group | Transplant With AKs; 5FU + PDT | Transplant With AKs; PDT Only | Normals With AKs; 5FU + PDT | Normals With AKs; PDT Only
Number analyzed (Participants) | 4 | 4 | 14 | 14
CR (% reduction)
  At 3 months post-PDT | 76.7 [46.1 to 100] | 34.6 [4.3 to 64.8] | 73.4 [64.0 to 82.7] | 49.5 [40.1 to 58.8]
  At 6 months post-PDT | 58.4 [26.3 to 90.4] | 23.8 [0 to 55.8] | 69.0 [55.1 to 82.9] | 43.1 [29.2 to 57.0]
  9 mos (see ClinCaRes2018)) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  12 mos (see ClinCaRes 2018) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Transplant With AKs; 5FU + PDT vs Transplant With AKs; PDT Only; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Normals With AKs; 5FU + PDT vs Normals With AKs; PDT Only; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Post Hoc Outcome: New AK Lesion Development
Description: The time (in months) following PDT treatment at which AK lesion counts first began to increase again. (Note: The nadir in AK lesion counts is reached at about 3 months in almost all patients).
Time Frame: 12 months post-PDT
Measure: Mean (Standard Deviation); unit: months
Groups:
- PDT Only: Patients who did not receive 5-FU prior to PDT
- 5-FU Followed by PDT: Patients who received a week of topical 5-FU pretreatment prior to PDT
Arm/Group | PDT Only | 5-FU Followed by PDT
Number analyzed (Participants) | 17 | 17
months | 8.1 (2.8) | 8.5 (2.4)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Solid Organ Transplant With AKs: Patients who have undergone kidney or liver transplant within 2 years and have at least 4 premalignant skin lesions on the face, ears, scalp, forearms and/or dorsal hands.
- Actinic Keratoses: Patients with at least 4 actinic keratoses on the face, ears, scalp, forearms and/or dorsal hands.
Arm/Group | Solid Organ Transplant With AKs | Actinic Keratoses
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/14
Other Adverse Events (participants affected / at risk) | 0/4 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Organ Transplant With AKs (N=4) | Actinic Keratoses (N=14)
Stroke (Vascular disorders) | 1 (1) | 0 (0) — Patient with lupus antioagulant, hospitalized for 2 transient ischemic attacks. Not thought to be related in any way to the skin photodynamic therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No